CLINICAL TRIAL: NCT04480567
Title: A Phase 1/2 Open-Label, Dose Escalation Study to Determine the Safety and Efficacy of BMN 307, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Phenylalanine Hydroxylase in Subjects with Phenylketonuria
Brief Title: AAV Gene Therapy Study for Subjects with PKU
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 307-201
Record Dates: First submitted 2020-07-08; First posted 2020-07-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; PAH Deficiency
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose 1 of BMN 307 (Experimental)
  Interventions: Drug: BMN 307
- Dose 2 of BMN 307 (Experimental)
  Interventions: Drug: BMN 307
- Dose 3 of BMN 307 (Experimental)
  Interventions: Drug: BMN 307

INTERVENTIONS:
Drug: BMN 307 — AAV Gene Therapy Infusion

SUMMARY:
This is a Phase 1/2, open-label, dose escalation study to evaluate the safety, efficacy and tolerability of BMN 307 in adult PKU subjects with PAH deficiency. Participants will receive a single administration of BMN 307 and will be followed for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with diagnosis of PKU which is a condition characterized by PAH deficiency
* Ability and willingness to maintain dietary protein intake consistent with baseline intake
* Willingness to abstain from hepatotoxic substances post-BMN 307 administration
* Willingness and capable per investigator opinion to comply with study procedures and requirements
* Willingness to use effective methods of contraception
* Plasma Phe levels > 600 µmol/L

Exclusion Criteria:

* Subjects with primary BH4 deficiency or other forms of BH4 metabolism deficiency
* Clinically significant liver dysfunction or disease
* Prior treatment with gene therapy
* Any condition that, in the opinion of the investigator or Sponsor, would prevent the subject from fully complying with the requirements of the study
* History of malignancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean Plasma Phe levels | baseline, week 12

SECONDARY OUTCOMES:
Change from baseline in mean Plasma Phe levels | baseline, week 96
Change from baseline in dietary protein intake from intact food | baseline, week 96
Number of participants with treatment-emergent adverse event | At 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (3):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Morristown Medical Center, Morristown, New Jersey
- University Hospital Birmingham NHS Foundation Trust, Birmingham, United Kingdom